CLINICAL TRIAL: NCT00886067
Title: An Open-label Positron Emission Tomography (PET) Study Using 2 [18F] F A85380 to Determine α4β2 Neuronal Nicotinic Receptor (NNR) Occupancy of AZD1446 After Oral Administration to Male and Non-fertile Female (Non-nicotine Users) Healthy Volunteers
Brief Title: Positron Emission Tomography (PET) Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: AstraZeneca
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D1950C00004; EudraCT No. 2008-008390-55
Record Dates: First submitted 2009-04-21; First posted 2009-04-22 (Estimated); Last update posted 2009-09-10 (Estimated); Status verified 2009-09

CONDITIONS: Healthy
Keywords: AZD1446; PET examination
MeSH Terms: interventions — 3-(5-chloro-2-furoyl)-3,7-diazabicyclo(3.3.0)octane; 2-fluoro-3-(2-azetidinylmethoxy)pyridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2-[18F]-F-A85380 (Experimental): Single microdose
  Interventions: Radiation: 2-[18F]-F-A85380
- AZD1446 (Experimental): Single oral administration
  Interventions: Drug: AZD1446

INTERVENTIONS:
Drug: AZD1446 — Solution, oral, single dose
  Arms: AZD1446
Radiation: 2-[18F]-F-A85380 — iv, single dose
  Arms: 2-[18F]-F-A85380

SUMMARY:
The primary purpose is to study the occupancy at the α4β2 neuronal nicotinic receptor's (NNRs) and to determine the relation between plasma concentration of AZD1446 and the occupancy at α4β2 NNRs.

ELIGIBILITY:
Inclusion Criteria:

* Physically healthy volunteers
* Body weight between 50 to 100 kg and body mass index (BMI) between 19 and 30 kg/m2

Exclusion Criteria:

* History of any clinically significant disease or disorder
* History of severe allergy/hypersensitivity reactions
* Participation in a PET examination as part of a scientific study during the past twelve months

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2009-04; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Determine whether and to what extent AZD1446 can displace radioligand 2-[18F]-F-A85380 from binding to α4β2 neuronal nicotinic receptors (NNRs) and to describe the relationship between plasma concentrations of AZD1446 and its occupancy at α4β2 NNRs. | One PET assessment on baseline day and one PET assessment at the drug treatment day
Plasma concentration (Cmax, tmax, AUC) | During time period of the PET assessment

SECONDARY OUTCOMES:
Safety and tolerability (AEs, vital signs, lab) | During the whole study

CONTACTS AND LOCATIONS:
Overall Officials: Björn Paulsson, MD, PhD, Study Director — AstraZeneca Södertälje; Ingemar, Bylesjö, MD, PhD, Principal Investigator — AstraZeneca CPU Huddinge
Locations (1):
- Research Site, Stockholm, Sweden